CLINICAL TRIAL: NCT02025166
Title: Comparison Between Two Analgesic Methods for Pain Relief Following Surgical Abortion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Lior Lowenstein, Gynecologist, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RMB343-13; RMB0343-13 (Other: Helsinki)
Record Dates: First submitted 2013-12-23; First posted 2013-12-31 (Estimated); Last update posted 2013-12-31 (Estimated); Status verified 2013-12

CONDITIONS: Pain
Keywords: Pain; abortion; paracetamol; lornoxicam
MeSH Terms: conditions — Pain | interventions — Acetaminophen; Analgesia; lornoxicam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paracetamol (Active Comparator): Pain treatment, aniline analgesics
  Interventions: Drug: Paracetamol; Drug: lornoxicam
- lornoxicam (Active Comparator): Pain treatment, nonsteroidal anti-inflammatory (NSAID)
  Interventions: Drug: Paracetamol; Drug: lornoxicam

INTERVENTIONS:
Drug: Paracetamol — Pain treatment with "aniline analgesics" (paracetamol) at the time of the procedure
  Other Names: Pain relief
Drug: lornoxicam — Pain treatment with "NSAID" (lornoxicam) at the time of the procedure
  Other Names: Pain relief

SUMMARY:
To compare between the efficacy of Paracetamol IV vs. Lornoxicam IV in pain relief following surgical abortion.

The medication will be given at the time of the procedure. Following the abortion, pain level will be evaluated.

DETAILED DESCRIPTION:
Patients with medical indication for surgical abortion during first trimester will be divided to two groups. The study groups, the surgeons and the nurses will be blinded to one of the treatment arms.

Pain will be evaluated at fixed intervals following the abortion. Comparison in pain levels between the study groups will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgical abortion for first trimester pregnancy

Exclusion Criteria:

* Chronic pelvic pain
* Fibromyalgia
* Pelvic inflammatory disease
* Chronic renal failure, liver disease, peptic ulcer
* cervical stenosis

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Pain | Two hours
  Pain level will be evaluated by VAS

CONTACTS AND LOCATIONS:
Overall Officials: Susana Mustafa, MD, Principal Investigator — Rambam Health Care Campus; Nibal Awad, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, Israel